CLINICAL TRIAL: NCT02137213
Title: Oral Naloxone for Treatment of Opioid-induced Constipation in Patients Receiving Methadone Maintenance Treatment
Brief Title: Feasibility Study of Oral Naloxone for Treatment of Methadone-induced Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Academic Health Science Centres (Other)
Responsible Party: Principal Investigator, Andriy V. Samokhvalov, MD, PhD, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 083/2013
Record Dates: First submitted 2014-05-12; First posted 2014-05-13 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Constipation
Keywords: Opioid-induced constipation; Methadone; Naloxone
MeSH Terms: conditions — Constipation; Opioid-Induced Constipation | interventions — Naloxone; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: Naloxone then placebo (Experimental): Subjects assigned to Arm A will receive methadone with naloxone for one week and then methadone with placebo for one week
  Interventions: Drug: Naloxone; Drug: Placebo
- Arm B: Placebo then naloxone (Experimental): Subjects assigned to Arm B will receive methadone with placebo for one week and then methadone with naloxone for one week
  Interventions: Drug: Naloxone; Drug: Placebo

INTERVENTIONS:
Drug: Naloxone — Naloxone will be added to oral methadone preparation in methadone:naloxone ratio of 50:1
  Other Names: Naloxone hydrochloride solution for injections 0.4 mg/ml
Drug: Placebo — Normal saline will be added to oral methadone preparations as placebo.
  Other Names: Bacteriostatic normal saline

SUMMARY:
At least 30% of patients receiving methadone maintenance therapy (MMT) are suffering from constipation that often affects effectiveness of MMT and increases its impact on health care system. Existing treatments include several over-the-counter medications which do not target the pathobiological basis of opioid-induced constipation and have limited effectiveness. At the same time well-known medication, naloxone, was already shown to help with constipation in patients receiving methadone for chronic pain, but was never tried in patients receiving methadone for opioid dependence. This study is aimed to try naloxone for treatment of opioid-induced constipation in MMT settings.

The investigators will enroll 20 patients receiving MMT and suffering from opioid-induced constipation. The study has a crossover design - all patients will receive one week of their regular methadone doses and one week of their regular methadone doses with naloxone added. Normal saline will be added to methadone-only formulations as placebo. Order of the weeks will be chosen randomly. Both subjects and investigators will be blinded to the study condition (i.e. whether naloxone or normal saline is added to methadone preparation on a given week).

Primary hypothesis: Patients receiving combination of oral methadone/naloxone in ratio 50:1 will have less severe symptoms of constipation compared to those receiving methadone only.

Secondary hypothesis: Addition of oral naloxone to methadone in a ratio 50:1 will not cause clinically significant opioid withdrawal symptoms.

DETAILED DESCRIPTION:
Background and rationale Opioid-induced constipation is the most common side effect of opioid therapy - depending on the settings up to 90% of patients taking opioids experience constipation with the most conservative estimate among MMT patients being 30%. Currently, the recommended treatment for opioid-induced constipation includes a combination of stool softeners, stimulants and osmotic laxatives - increased gastrointestinal secretions result in increased volume and softness of fecal masses, and more intense peristalsis promotes bowel voiding. The effectiveness of existing treatments for opioid-induced constipation is limited - they are effective in approximately 50% of cases, often have side effects such as abdominal cramping and diarrhea and, most importantly, do not address the pathobiological basis of opioid-induced constipation. Opioids in general and methadone in particular act on peripheral opioid receptors located in myenteric and submucosal plexus and cause relaxation of longitudinal and increased tone of inner circular smooth muscles as well as decreased gastrointestinal secretions that in turn result in constipation. The most logical therapeutic approach to the treatment of opioid-induced constipation in MMT would be using opioids that cause selective local reversal of μ-opioid activation with a peripherally-acting opioid antagonist such as naloxone, which when administered orally does not have systemic effects due to extremely low oral bioavailability.

Objectives The primary objective is to evaluate the effectiveness of a combination of methadone and naloxone in 50:1 for treatment of opioid-induced constipation in MMT patients. The secondary objective of the study is to assess the likelihood of development of opioid withdrawal symptoms in MMT patients who receive combination of methadone and naloxone compared to those who receive methadone only.

Design Study has a double-blind placebo-controlled crossover design: following signing informed consent and initial assessment 20 subjects who meet eligibility criteria will be randomized into one of two groups: group A will receive combination of methadone and naloxone in a ratio of 50:1 shown to be safe and effective in other trials during week 1 of the study and methadone only during week 2 of the study. Group B will receive methadone only during week 1 of the study and combination of methadone and naloxone in a ratio of 50:1 during week 2 of the study. Thus, all participants will receive combination of methadone and naloxone for one week and methadone alone for one week. Neither study participants, nor the pharmacists observing the doses, nor study personnel will know if naloxone is added to subjects' methadone preparations. Allocation to Group A or Group B will be done by random assignment. The pharmacy research medication management service will prepare the randomization code such that there will be a balanced assignment after every 4 subjects. Bowel functioning will be assessed quantitatively primarily using the Bowel Function Index (BFI) at initial assessment and at the end of weeks one (day 8) and two of the study (day 15). Also data on the number of complete spontaneous bowel movements (CSBMs), their temporal relationship to medication administration and outcome will be collected every day prior to administration of the next dose of methadone. In addition to parameters of bowel functioning Subjective Opiate Withdrawal Scale (SOWS) will be administered daily in order to assess potential opioid withdrawal symptoms.

Statistical Methods/Data Analysis Primary endpoint of the study is the reduction of constipation symptoms severity as measured by the difference between BFI scores taken after one week of receiving combination of methadone and naloxone and after one week of receiving methadone only. Secondary endpoint of the study is the occurrence of opioid withdrawal symptoms as measured by the difference between the mean SOWS scores taken daily during each of two weeks of the study. Paired t-test will be used to compare BFI and mean number of CSBMs between the weeks of treatment with a combination of methadone and naloxone and methadone alone as well as to compare average SOWS scores between the weeks of treatment with a combination of methadone and naloxone and methadone alone.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* must be a registered CAMH methadone maintenance program client
* must be in a maintenance stage of MMT program (at least 6 weeks in MMT)
* stable methadone dose taken once daily (no methadone dose change in the past 4 weeks)
* methadone dose between 20 mg and 140 mg/day (normal range of methadone doses prescribed in CAMH opioid dependence clinic)
* Bowel Functioning Index score ≥ 30 (reference range for non-constipated patients is 0-28.8)
* less than 3 bowel movements in the week prior to initiation

Exclusion Criteria:

* patients prescribed opioids other than methadone
* patients who use opioids recreationally
* patients prescribed methadone for pain management
* patients receiving methadone in split doses
* pregnancy
* allergy or sensitivity to naloxone
* current gastrointestinal disorder (chronic colitis, Crohn disease etc.)
* taking medications with known strong anticholinergic effects (e.g. amitryptiline)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Severity of constipation symptoms | One week
  Severity of constipation symptoms will be measured after one week of receiving methadone with naloxone and after one week of receiving methadone alone in both arms of the study.

SECONDARY OUTCOMES:
Severity of opioid withdrawal symptoms | Two weeks
  The severity of opioid withdrawal symptoms will be assessed using Subjective Opioid Withdrawal Scale (SOWS) over the course of the study (2 weeks for each participant)

CONTACTS AND LOCATIONS:
Overall Officials: Andriy V Samokhvalov, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre. — http://www.camh.ca/en/research